CLINICAL TRIAL: NCT00272194
Title: The Ambu® Laryngeal Mask as an Intubation Conduit For Patients Undergoing Routine General Anesthesia
Brief Title: Ambu® Laryngeal Mask as an Intubation Conduit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Carin A. Hagberg, Professor and Chairman, Joseph C. Gable, M.D., Endowed Chair, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HSC-MS-05-0347
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Intubation, Endotracheal
Keywords: Endotracheal Intubation; Supraglottic Airway
MeSH Terms: interventions — Laryngeal Masks

INTERVENTIONS:
Device: Ambu Laryngeal Mask
Device: Aintree Exchange Catheter
Device: Laryngeal Mask Airway

SUMMARY:
The purpose of this study is to determine if the Ambu Laryngeal Mask can be used as an intubation conduit for endotracheal intubation.

DETAILED DESCRIPTION:
The laryngeal mask airway (LMA) is an established supra-glottic device that provides better ventilation than traditional mask ventilation and is less invasive than endotracheal intubation. Being less invasive, it is commonly used for short elective surgical procedures. Its ability to be both easily and rapidly inserted also makes it useful as a rescue device in difficult and failed intubations. Being a supra-glottic device, the LMA does not protect patients from regurgitation and aspiration. Additionally, patients requiring alternative positions, such as prone or lateral, or those having surgery in the neck/head area are contra-indicated for LMA use due to risk of possible movement of the LMA, and therefore possible loss of airway patency. Thus, the LMA can be utilized as an intermediary method of airway management to endotracheal intubation.

The manufacturer of the reusable LMA-ClassicTM states that "the success rate of intubation through the standard LMA-ClassicTM is highly variable (30-93%)," whereas the success rate of the disposable version, LMA-UniqueTM, has been found to be only 21%1. An LMA specifically designed for intubation now exists and improves the success rate of intubation. The reusable LMA-FastrachTM or Intubating-LMATM (ILMA) is a rigid and anatomically curved airway tube. It is wide enough to accommodate 8.0 mm cuffed endotracheal tubes. Attached to the ILMA is a rigid handle to aid in one-handed insertion, removal, and adjustment. Success rates for intubating through the ILMA are 96.5% when inserted blindly and 100% with fiberoptic guidance2. No disposable version of the ILMA presently exists.

The Ambu® Laryngeal Mask (ALMA) is a new disposable laryngeal mask with an anatomical curve similar to the ILMA. The reasons for the use of disposable products can be many and varied. The residual risk of the transmission of germs and protein particles represents one indication. If supra-glottic airway devices are used electively or in emergencies, e.g. for HIV-positive patients or those infected with Creutzfeldt-Jacob disease, reuse of the products is not desirable. Disposable products, on the other hand, offer the benefit that the transmission of germs is avoided, and at the same time offer considerable economic advantages due to the much lower price of the product. The disposable ALMA has been proven as an effective and safe supra-glottic airway device3. Upon fiberoptic visualization through its shaft, the glottis was visualized 91.5% of the time, indicating that this device may be used as an intubation conduit. The purpose of this study is to determine if the ALMA is also safe and effective as an intubating conduit. The hypothesis is that the ALMA will perform as well as, if not better than the LMA-UniqueTM.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ASA 1-3 presenting for an elective surgical procedure
* The patient is 18-65 years of age
* The patient weighs > 50 kg with a BMI < 30 kg/m2
* The patient has a Mallampati grade I -III airway
* The patient is undergoing general anesthesia with controlled ventilation for minor routine surgical procedures
* The period of anesthesia time is >30 minutes

Exclusion Criteria:

* The patient is an ASA classification 4
* The patient is < 18 or >65 years of age
* The patient weighs < 50 kg or has a BMI > 30 kg/m2
* The patient has a history of inadequate cervical mobility
* The patient has a history or signs of difficult airway management
* The patient has a Mallampati grade IV Class airway
* The patient has a mouth opening < 2.5 cm
* The patient has an oral cavity disease
* The patient has a cervical malformation
* The patient had upper respiratory tract symptoms in the previous 10 days
* The patient is to have surgery performed to the head/neck or thoracoabdominal cavities needing to be paralyzed, or in the lateral/prone position
* The patient is considered at risk of aspiration (non-fasted, gastroesophageal reflux/disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time and number of attempts required; Level of difficulty; Degree of irritation of the pharynx, epiglottis, and arytenoids

SECONDARY OUTCOMES:
vital signs, oxygen saturation, end-tidal carbon dioxide

CONTACTS AND LOCATIONS:
Overall Officials: Carin A. Hagberg, M.D., Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States